CLINICAL TRIAL: NCT00276588
Title: Phase II Trial of Gemcitabine/Paraplatin® (Carboplatin) Followed by Taxol® (Paclitaxel) in Patients With Performance Status = 2,3 or Other Significant Co-Morbidity (HIV Infection or s/p Organ Transplantation) in Advanced Non-Small Cell Lung Cancer
Brief Title: Gemcitabine and Carboplatin Followed by Paclitaxel in Treating Patients With Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: JHOC-J0428, CDR0000450843; P30CA006973 (NIH); JHOC-J0428; BMS-JHOC-J0428; JHOC-BRAAN-21048; MSGCC-0060; JHOC-04112308
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2010-08

CONDITIONS: Lung Cancer
Keywords: adenocarcinoma of the lung; adenosquamous cell lung cancer; large cell lung cancer; recurrent non-small cell lung cancer; squamous cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Gemcitabine; Paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: gemcitabine hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, carboplatin, and paclitaxel work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with carboplatin followed by paclitaxel works in treating patients with stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy and tolerability of gemcitabine hydrochloride and carboplatin followed by paclitaxel in patients with stage IIIB-IV non-small cell lung cancer in regard to response rate, median survival, and one year survival.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is multicenter study.

* Part 1: Patients receive carboplatin IV over 30 minutes on day 1 and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 3 weeks for 2 courses. In week 7, all patients proceed to part 2 regardless of disease response.
* Part 2: Patients receive paclitaxel IV over 1-3 hours once weekly for 6 weeks. Treatment repeats every 8 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 46 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small lung cancer (NSCLC) of any of the following histologic types:

  * Squamous cell
  * Adenocarcinoma
  * Large cell carcinoma
  * Unspecified
* Evidence of at least 1 of the following criteria:

  * Newly diagnosed inoperable stage IIIB (pleural effusion) disease
  * Patients with stage III disease who are unable to undergo combined modality therapy
  * Stage IV disease
  * Recurrent non-small cell lung cancer regardless of site
  * Diagnosis based on sputum cytology acceptable if confirmed by an independent pathologic review
* Patients must have measurable or evaluable disease

  * Measurable or evaluable disease must be outside the previous radiation field or a new lesion must be present
* Patients with brain metastases are eligible, provided they are either asymptomatic (no neurological symptoms or signs, no evidence of midline shift), or controlled (i.e., after surgical resection or radiotherapy/radiosurgery), and off all steroid therapy for at least two weeks with no evidence of progression by symptoms or radiologic imaging

PATIENT CHARACTERISTICS:

* ECOG performance status of 2 or 3 OR HIV-positive OR underwent prior status post organ transplantation
* No active serious infection (except for HIV infection)
* No symptomatic, untreated malignant pericardial effusion
* No congestive heart failure
* No other serious underlying medical condition that would otherwise impair their ability to receive protocol treatment
* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm ^3
* Creatinine clearance ≥ 40 mL/min
* Creatinine ≤ 1.8 mg/dL
* Bilirubin < 1.5 mg/dL
* SGOT ≤ 2 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Males or females of reproductive potential may not participate unless they have agreed to use effective barrier contraceptive methods
* No prior malignancy within the past 5 years except for adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior chemotherapy is not allowed
* At least three weeks since prior radiotherapy and recovered from all toxicities
* At least three weeks must have elapsed from major surgery and recovered from all adverse effects of surgery
* No prior colony-stimulating factors or interferon
* No concurrent hormonal, biologic, or radiotherapy to measurable lesions

  * Patients may receive concurrent palliative radiotherapy to small-field nonmeasurable sites of disease (e.g., painful bony metastases)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2005-07; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Overall survival
Progression-free survival
Time to treatment failure
Time to progression

SECONDARY OUTCOMES:
Duration of response (complete response and partial response)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Brahmer, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland

REFERENCES:
- [Result] Bridges BB, Thomas L, Hausner PF, Doyle LA, Bedor M, Smith R, Brahmer J, Edelman MJ. Phase II trial of gemcitabine/carboplatin followed by paclitaxel in patients with performance status=2,3 or other significant co-morbidity (HIV infection or s/p organ transplantation) in advanced non-small cell lung cancer. Lung Cancer. 2008 Jul;61(1):61-6. doi: 10.1016/j.lungcan.2007.11.009. Epub 2008 Jan 16. PMID 18201795